CLINICAL TRIAL: NCT03800875
Title: A Randomized, Controlled, Crossover Trial to Assess a Dual-hormone (Insulin-pramlintide) Closed-loop Delivery Without Carbohydrate Counting in Regulating Glucose Levels in Adults With Type 1 Diabetes
Brief Title: Insulin-plus-pramlintide Closed-loop Strategy to Regulate Glucose Levels Without Carbohydrate Counting
Acronym: Dual
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Diabetes Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Triple Hormone
Record Dates: First submitted 2018-06-27; First posted 2019-01-11 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Pramlintide; Insulin; Dual-Hormone; Closed-Loop; Artificial Pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Insulin-Pramlintide Closed-Loop Strategy (Experimental): Fast-acting insulin will be delivered using two separate infusion pumps. The pumps' infusion rates will then be changed manually based on the computer-generated recommendation. The computer-generated recommendations are based on a dosing algorithm. With no-meal announcement or carbohydrate counting, the dual-hormone closed-loop system will be fully reactive, and insulin and pramlintide dosages will be based solely on sensor readings
  Interventions: Drug: 27-hour inpatient intervention
- Insulin-alone Closed Loop Strategy (Active Comparator): Fast-acting insulin will be delivered by a subcutaneous insulin infusion pump based on an algorithm that automatically adjusts insulin rates based on a dosing algorithm. The carbohydrate content for every ingested meal will be entered into the algorithm to calculate the insulin prandial bolus based on each participant's insulin-to-carbohydrate ratio. The carbohydrate content will be entered at the onset of the meal.
  Drug(s): Insulin (FiAsp)
  Interventions: Drug: 27-hour inpatient intervention

INTERVENTIONS:
Drug: 27-hour inpatient intervention — Subjects will be admitted at the research facility at 19:00. Each 27-hour intervention visit includes 3 standardized meals (8:00, 12:00, and 17:00), an evening snack (22:00) and an overnight stay. The glucose level as measured by the real time sensor will be entered manually into the computer every 10 minutes. The infusion rate of either insulin alone or insulin and pramlintide will be changed manually based on the computer generated recommendation. The computer generated recommendations are based on a predictive algorithm.

SUMMARY:
Closed-loop system systems that are shown to alleviate the burden of carbohydrate counting without degrading glucose control are still lacking. In this proposal, the investigators aim to develop a novel, fully-automated, closed-loop system that delivers insulin and pramlintide that controls postprandial glucose levels without any input from the user.

DETAILED DESCRIPTION:
Meal carbohydrate content is the main determinant of prandial insulin needs, and consequently, accurate carbohydrate counting is recommended for type 1 diabetes. Advances in glucose sensors have motivated the development of the closed-loop system to automatically regulate glucose levels in individuals with type 1 diabetes. In the closed-loop system, a dosing algorithm adjusts the pump insulin infusion rate based on continuous glucose sensor readings.

Closed-loop system systems that are shown to alleviate the burden of carbohydrate counting without degrading glucose control are still lacking. In this proposal, the investigators aim to develop a novel, fully-automated, closed-loop system that delivers insulin and pramlintide that controls postprandial glucose levels without any input from the user. Thus, the two hormones' role in the postprandial state will be as follows:

1. Insulin: to reduce plasma glucose levels. Insulin delivery needs to be aggressive to counter-act fast increase in post-meal glucose levels.
2. Pramlintide: to slow gastric emptying and aim insulin in efficiently controlling postprandial glucose levels.

The aim of this study is to assess a fully automated, dual-hormone, closed-loop system that delivers insulin, and pramlintide to control glucose levels without degrading overall glycemic control compared to an insulin-alone closed-loop system with carbohydrate-matched boluses.

The investigators hypothesize that the dual-hormone closed-loop system will alleviate carbohydrate-counting burden (fully reactive system) without degrading glucose control compared to the insulin-alone closed-loop system.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of age.
2. Clinical diagnosis of type 1 diabetes for at least 12 months. The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.
3. Insulin pump therapy for at least 6 months.
4. HbA1c ≤ 12% in the last 6 months.

Exclusion Criteria:

1. Current or ≤ 1 month use of other antihyperglycemic agents (SGLT2, GLP-1, Metformin, Acarbose, etc.…).
2. Severe hypoglycemic episode within one month of admission.
3. Severe diabetic ketoacidosis episode within one month of admission.
4. Pregnancy.
5. Known or suspected allergy to the study drugs.
6. Gastroparesis.
7. Use of prokinetic drugs that stimulate gastric emptying (domperidone, cisapride, metoclopramide).
8. Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator.
9. Recent (< 6 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
10. Current use of glucocorticoid medication.
11. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
12. Failure to comply with team's recommendations (e.g. not willing to eat meals/snacks, not willing to change pump parameters, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2020-09-19 (Actual); Study Completion 2020-09-19 (Actual)

PRIMARY OUTCOMES:
Total percentage of time (22:00-22:00) that the glucose concentration remained within 3.9 and 10.0 mmol/L | 24 hours

SECONDARY OUTCOMES:
Total percentage of time (22:00-22:00) that the glucose concentration remained within specified ranges. | 24 hours
  a. between 3.9 and 7.8 mmol/L; b. below 3.9 mmol/L; c. between 3.9 and 10 mmol/L d. below 3.3 mmol/L; e. below 2.8 mmol/L; f. above 7.8 mmol/L; g. above 10 mmol/L; h. above 13.9 mmol/L; i. above 16.7 mmol/L.
Percentage of overnight time (24:00-8:00) that the glucose concentration remained within specified ranges. | 8 hours
  a. between 3.9 and 7.8 mmol/L; b. between 3.9 and 10 mmol/L; c. below 3.9 mmol/L; d. below 3.3 mmol/L; e. below 2.8 mmol/L; f. above 7.8 mmol/L; g. above 10 mmol/L; h. above 13.9 mmol/L; i. above 16.7 mmol/L.
Total amount of insulin delivered to the participant | 24 hours
Mean sensor glucose concentration during the overnight stay | 8 hours
Number of participants experiencing hypoglycemia requiring oral treatment during: a. the overall study period; b. the night; c. the day | 27 hours
The number and severity of gastrointestinal sysmptoms experienced by a participant | 27 hours
  GI symptoms include: nausea, vomiting, bloating and heartburn
Mean daytime insulin concentration | 14 hours
Mean daytime concentration of amylin | 14 hours
Total amount of pramlintide delivered to the participant | 24 hours
Mean glucose level | 24-hour period

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tsoukas, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The raw data (i.e., insulin delivery, glucose levels, individual participant data) and informed consent form could be shared by the corresponding author, ahmad.haidar@mcgill.ca, upon reasonable request for academic purposes, subject to Material Transfer Agreement and approval of McGill University Health Center's Research Ethics Board. All data shared will be de-identified. The study protocol will be available with publication.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] Tsoukas MA, Majdpour D, Yale JF, Fathi AE, Garfield N, Rutkowski J, Rene J, Legault L, Haidar A. A fully artificial pancreas versus a hybrid artificial pancreas for type 1 diabetes: a single-centre, open-label, randomised controlled, crossover, non-inferiority trial. Lancet Digit Health. 2021 Nov;3(11):e723-e732. doi: 10.1016/S2589-7500(21)00139-4. Epub 2021 Sep 24. PMID 34580055